CLINICAL TRIAL: NCT01500070
Title: PREVENT: a Prospective, Multi-center, Monitored Trial Investigating the Implant of the Promus Everolimus-Eluting Stent System in Critically Ischemic Lesions BTK
Brief Title: PREVENT: Promus BTK
Acronym: PREVENT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Flanders Medical Research Program (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRP-101020
Record Dates: First submitted 2011-12-19; First posted 2011-12-26 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Claudication; Drug-Eluting Stent; BTK; Everolimus; CLI
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug-eluting stent (Experimental): Patients implanted with the PROMUS ELEMENT Everolimus-Eluting Stent System (Boston Scientific) or the PROMUS ELEMENT PLUS Everolimus-Eluting Stent System (Boston Scientific).
  Interventions: Device: Everolimus-Eluting Stent (PROMUS ELEMENT)

INTERVENTIONS:
Device: Everolimus-Eluting Stent (PROMUS ELEMENT) — PROMUS ELEMENT Everolimus-Eluting Stent System (Boston Scientific) or PROMUS ELEMENT PLUS Everolimus-Eluting Stent System (Boston Scientific).

SUMMARY:
This is a single-arm, prospective, multi-center monitored trial recruiting patients with critical limb ischemia and with one or more lesions in the arteries below the knee. The immediate and long-term (up to 12 months) outcome of the PROMUS ELEMENT Everolimus-Eluting Stent System (Boston Scientific) and the PROMUS ELEMENT PLUS Everolimus-Eluting Stent System (Boston Scientific) will be evaluated.

In 2 Belgian centers, 3 German centers and 1 New Zealand center a total of 70 patients will be recruited. Primary endpoint is primary patency at 12 months, defined as absence of restenosis (≥50% stenosis) or occlusion within the originally treated lesion based on angiography.

ELIGIBILITY:
General Inclusion Criteria:

* Patient presenting with rest pain or minor tissue loss (Rutherford class 4 or 5)
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient is >18 years old
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study
* Patient has a projected life-expectancy of at least 12 months
* The treating physician consider the patient eligible for below-the-knee treatment with the PROMUS ELEMENT Stent (Boston Scientific) and PROMUS ELEMENT PLUS Stent (Boston Scientific)
* Male, infertile female, or female of child bearing potential practicing an acceptable method of birth control with a negative pregnancy test within 7 days prior to study procedure

Angiographic Inclusion Criteria:

* Single or multiple lesions with minimally 70% stenosis in one or more infrapopliteal arteries, including the tibiofibular trunk
* A maximum of two focal target lesions in one or more infrapopliteal vessels
* Length of lesion is maximally 40 mm, allowing maximally 2 planned stents to be implanted
* Target vessel diameter visually estimated to be >2.5mm and <4.0mm
* Guidewire and delivery system successfully traversed lesion

General Exclusion Criteria:

* Patient refusing treatment
* Previously implanted stent in the artery to be treated
* Failed PTA of target lesion/vessel less than 3 months prior to study procedure
* The reference segment diameter is not suitable for the available stent design
* Untreated flow-limiting inflow lesions
* Perioperative unsuccessful ipsilateral percutaneous vascular procedure to treat inflow disease just prior to enrollment
* Any previous surgery in the target vessel (including prior ipsilateral crural bypass)
* Aneurysm in the target vessel
* Patient presents with renal failure, evidenced by a serum creatinine level >2.0mg/dL
* Patient presents with platelet levels above or below normal range
* Non-atherosclerothic disease resulting in occlusion (e.g. embolism, Buerger's disease, vasculitis)
* Severe medical comorbidities (untreated CAD/CHF, severe COPD, metastatic malignancy, dementia, etc) or other medical condition that would preclude compliance with the study protocol or 1-year life expectancy
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Any previously known coagulation disorder, including hypercoagulability
* Contraindication to anticoagulation or antiplatelet therapy
* Known allergies to stent or stent components
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* Patient with known hypersensitivity to heparin, including those patients who have had a previous incidence of heparin-induced thrombocytopenia (HIT) type II
* Currently participating in another clinical research trial
* Angiographic evidence of intra-arterial thrombus or atheroembolism from inflow treatment
* Target lesion access not performed by transfemoral approach.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Absence of restenosis (50% stenosis) or occlusion within the originally treated lesion based on angiography.

SECONDARY OUTCOMES:
Technical success | 1 day post-procedure
  The ability to cross and dilate the lesion to achieve residual angiographic stenosis no greater than 30%.
Hemodynamic primary patency rate | 1, 6 and 12 month follow-up
  Patients that present without a hemodynamically significant stenosis at the target area on duplex ultrasound (systolic velocity ratio no greater than 2.4) and without prior TLR are defined as being primary patent at the given follow-up.
Limb-salvage | 1, 6 and 12 month follow-up
  Absence of major amputation, defined as amputation at or above the ankle, as opposed to minor amputation, being an amputation at or below metatarsal level, preserving functionality of the foot).
Primary assisted patency rate | 1, 6 and 12 month follow-up
  Defined as flow through the treated lesion maintained by repeat percutaneous intervention completed prior to complete vessel closure.
Secondary patency rate | 1, 6 and 12 month follow-up
  Defined as flow through the treated lesion maintained by repeat percutaneous intervention after occlusion of the target lesion.
Target lesion revascularization (TLR) | 1 day, 1 month, 6 month and 12 month follow-up
  Defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5 mm proximal and distal to the treated lesion edge.
Clinical success at follow-up | 1 day, 1 month, 6 month and 12 month follow-up
  Defined as an improvement of Rutherford classification at 1 day and 1, 6, 12-month follow-up of one class or more as compared to the pre-procedure Rutherford classification.
Improvement of ankle-brachial index (ABI) | 1 day, 1 month, 6 month and 12 month follow-up
  Defined as an increase of the ABI at 1 day and 1, 6, 12-month follow-up compared to baseline in subjects with compressible arteries and baseline ABI <0.9.
Serious Adverse Events (SAE) | 1 day, 1 month, 6 month and 12 month follow-up
  Defined as any clinical event that is fatal, life-threatening, or judged to be severe by the investigator; resulted in persistent or significant disability; necessitated surgical or percutaneous intervention; or required prolonged hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bosiers, MD, Principal Investigator — AZ Sint Blasius, Dendermonde, Belgium
Locations (8):
- Belgium (4):
  - Imelda Hospital, Bonheiden, Antwerpen
  - OLV Aalst, Aalst, Oost-Vlaanderen
  - AZ Sint-Blasius, Dendermonde, Oost-Vlaanderen
  - RZ Heilig Hart Tienen, Tienen
- Germany (3):
  - Herzzentrum Bad-Krözingen, Bad-Krözingen, Land Baden-Württemberg
  - St. Fransiskus Hospital, Münster, North Rhine-Westphalia
  - Herzzentrum Leipzig, Leipzig, Saxony
- Auckland City Hospital, Auckland, Auckland, New Zealand